CLINICAL TRIAL: NCT01434277
Title: A Single-Center Study Evaluating the Safety of a New Preservative in an OTC Lubricant Eye Drop Used QID in Healthy Adults and in Subjects Diagnosed With Dry Eye
Brief Title: Safety Evaluation of a New Preservative in a Lubricating Eye Drop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: UNKEDI0003
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Dry Eye Syndromes
Keywords: Preservative; Eye Drops
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Subjects (Experimental): Healthy Subjects instill 1-2 drops of the experimental eye drops into each eye four times per day for two weeks.
  Interventions: Other: Eye Drops with Experimental Preservative
- Dry-Eye Subjects (Experimental): Dry-Eye Subjects instill 1-2 drops of the experimental eye drops into each eye four times per day for two weeks.
  Interventions: Other: Eye Drops with Experimental Preservative

INTERVENTIONS:
Other: Eye Drops with Experimental Preservative — Glycerin, Hypromellose, Polyethylene glycol 400 with experimental preservative PQ-42
  Other Names: PF-006676

SUMMARY:
This study is to evaluate the safety of a new preservative in a lubricant eye drop used four times a day in healthy adults and subjects diagnosed with dry eye.

DETAILED DESCRIPTION:
Single-site, open-labeled study. Twenty two subjects will be enrolled into the healthy adult group and twenty two subjects into the dry eye group. Each subject will be in the study for approximately 2 weeks (treatment) and seen at three study Visits: Visit 1 (Day 0, Baseline), Visit 2 (Day 7 +/- 1) and Visit 3 (Day 14 +/- 1). Dosing regimen is 1-2 drops into each eye, four times daily, for two weeks. Assessments will be comprised of visual acuity, slit lamp biomicroscopy, fluorescein corneal staining, and product comfort.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able to follow all study instructions and attend all required study visits
* Provide written informed consent
* Visual health and eye comfort within protocol-specified parameters
* Women of child-bearing potential must have a negative urine pregnancy test at screening, not be breast-feeding, and agree to use a protocol-specified acceptable form of birth control throughout the study

Exclusion Criteria:

* Any medical condition or history, or ocular scores, or use of any drug, device or medication that, per protocol or in the opinion of the investigator, might compromise the safety of the subject or analysis of the study results.
* Use of contact lenses outside protocol allowance
* Self-reported pregnancy, positive urine pregnancy test, breast-feeding; intends to become pregnant or breast-feed during the duration of the study, refuses protocol-specified urine pregnancy testing, and/or does not use protocol-specified birth control methods and agree to continue doing so for the duration of the study.
* Participated in an investigational drug or device trial within 30 days of entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Post-dose Product Comfort | baseline, Within Two weeks
  Product (ocular) comfort was assessed for each eye immediately, and at 1, 2, and 3 minutes following dosing at Visit 1 and 3 using a scale ranging from 0 to 10, where 0 is very uncomfortable and 10 is very comfortable.
Change from Baseline in Pre-Dose Visual Acuity | baseline, Within Two weeks
  Change from Baseline in Pre-Treatment Means of Pre-Dose Visual Acuity on the LogMAR scale. (The LogMAR scale converts the geometric sequence of a traditional chart to a linear scale. It measures visual acuity loss; positive values indicate vision loss, while negative values denote normal or better visual acuity.)
Change from Baseline in Pre-dose Inferior Staining | baseline, Within Two weeks
  Means and Differences from Visit 1 in Pre-Dose Inferior Staining
Change from Baseline in Mean Corneal Staining | baseline, Within Two Weeks
  Mean Corneal Staining averaging over the 5 corneal regions and averaging over both eyes (NEI scale 0-3)
Change from Baseline in Pre-Dose Central Staining | baseline, Within Two Weeks
  Pre-dose Central Staining: Means and Differences from Visit 1
Change from Baseline in Pre-Dose Superior Staining | baseline, Within Two Weeks
  Pre-Dose Superior Staining: Means and Differences from Visit 1
Change from Baseline in Pre-Dose Temporal Staining | baseline, Within Two Weeks
  Pre-dose Temporal Staining: Means and Differences from Visit 1
Change from Baseline in Pre-Dose Nasal Staining | baseline, Within Two Weeks
  Pre-dose Nasal Staining: Means and Differences from Visit 1
Change from Baseline in Pre-Dose Average Staining | baseline, Within Two Weeks
  Pre-dose Average Staining: Means and Differences from Visit 1
Changes in Slit-Lamp Findings: Eye Structure: Lid | Within Two Weeks
  Slit-lamp findings were recorded for the Lid ocular structure at 6 time points
Changes in Slit-Lamp Findings: Eye Structure: Lens | baseline, Within Two Weeks
  Slit-lamp findings were recorded for the Lens ocular structure at 6 time points
Changes in Slit-Lamp Findings: Eye Structure: Conjunctiva | baseline, Within Two Weeks
  Slit-lamp findings were recorded for the Conjunctiva ocular structure at 6 time points
Change from Baseline in Slit-Lamp Findings: Eye Structure: Cornea | baseline, Within Two Weeks
  Slit-lamp findings were recorded for the Cornea ocular structure at 6 time points

CONTACTS AND LOCATIONS:
Overall Officials: Sherryl Frisch, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- ORA, Inc., Andover, Massachusetts, United States